CLINICAL TRIAL: NCT02161289
Title: Behavioral and Biomedical HIV Prevention Interventions for Thai Men Who Have Sex With Men.
Acronym: HIV-NAT 120
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: The HIV Netherlands Australia Thailand Research Collaboration (Other); Johns Hopkins University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 120
Record Dates: First submitted 2014-05-28; First posted 2014-06-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: HIV Testing, MSM
Keywords: 100 HIV-negagtve MSM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives

1. To evaluate the acceptability and feasibility of "standard HIV prevention package" among Thai men who have sex with men (MSM)
2. To conduct a pilot study to demonstrate the acceptability and feasibility of internet-based social networking, asymptomatic sexually transmitted infection diagnosis and treatment and pre-exposure prophylaxis strategies as "potential HIV prevention methods" among Thai MSM
3. To use mathematical modeling to identify the most effective HIV prevention package optimized for Thai MSM

Subject population: HIV-negative MSM clients of the Thai Red Cross Anonymous Clinic (TRC-AC), age ≥18 years old,Each participant will have a 12-month follow-up duration in the study.

DETAILED DESCRIPTION:
Study design and methodology:

We will conduct a pilot study among 100 MSM participants who will be enrolled from the TRC-AC and will be followed up for 12 months. Participants will be followed at baseline, months 1 and 3, and then every 3 months. Interventions in the "standard HIV prevention package" to be provided at every clinic visit include anti-HIV testing, risk reduction counseling, provisions of free condoms and lubricants and diagnosis and treatment of symptomatic sexually transmitted infections (STI). All participants will also have access to non-occupational post-exposure prophylaxis (nPEP) without charge as part of the standard HIV prevention package. In addition, we will test for acceptability and feasibility of the "potential HIV prevention methods" which include:

1) Internet-based social networking to distribute and stimulate discussion of HIV prevention information (2) Asymptomatic STI diagnosis and treatment for every participant at baseline visit and every 6 months (3) Oral and topical pre-exposure prophylaxis (PrEP) strategies using placebo tablet and gel.

The meta-analysis of various behavioral and biomedical HIV prevention studies among MSM will be done in parallel with the pilot study in order to gather information for mathematical modeling and finally to inform the design of a larger study. Data acquired from the pilot study will be used for mathematical modeling of HIV transmission among MSM. The output from the modeling will directly inform HIV preventative interventions to be evaluated empirically among MSM in Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or older
2. Have documented negative HIV EIA or CMIA test at screening
3. Live in or near Bangkok
4. Have a history of anal sex with men
5. Understand the study and sign informed consent form.

Exclusion Criteria:

1. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with ability to give informed consent
2. Persons with history of urinary tract stone

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men who have sex with men in Thailand
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Acceptability | 12 month
  An intervention will be defined as acceptable if the uptake is at least 60%.
Feasibility | 12 months
  Feasibility endpoints will be a combination of the ability to recruit subjects, subjects' adherence to each HIV prevention methods, ability for staff to perform procedures according to the protocol and an overall lost to follow up rate of 5% or less per year.

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathumwan,, Bangkok, Thailand